CLINICAL TRIAL: NCT05287529
Title: Telehealth Delivery of the Yoga for Seniors Program
Brief Title: In-home Yoga for Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1278; A176000 (Other: UW Madison); Protocol Approved 10/20/2021 (Other: UW Madison); ICTR Pilot (Other Grant/Funding Number: UWF Wisconsin Partnership)
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Aging Well
Keywords: underserved populations; yoga; elderly; movement; activity; balance; social isolation; falls
MeSH Terms: conditions — Motor Activity; Social Isolation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-Week Yoga Class (Experimental): Randomized to immediately begin an 8-week Yoga Class via Telehealth
  Interventions: Behavioral: Yoga Via Telehealth - Immediately
- Waitlisted for 8-Week Yoga Class (Active Comparator): Randomized to start an 8-week Yoga Class via Telehealth 8-weeks from the start of the study.
  Interventions: Behavioral: Yoga Via Telehealth - Waitlisted

INTERVENTIONS:
Behavioral: Yoga Via Telehealth - Immediately — The yoga program is an in-home, chair-assisted yoga class focused on balance. Each class will be led by a certified yoga teacher who has completed training the the yoga for Seniors Program. Classes will consist of no more than 12 participants. Each class will be attended by a local community member who will facilitate community building before and after class and will be available to activate local emergency medical services in the unlikely event that the need arises. Classes are 75 minutes in duration and meet two times per week.
  Arms: 8-Week Yoga Class
Behavioral: Yoga Via Telehealth - Waitlisted — The yoga program is an in-home, chair-assisted yoga class focused on balance. Each class will be led by a certified yoga teacher who has completed training the the yoga for Seniors Program. Classes will consist of no more than 12 participants. Each class will be attended by a local community member who will facilitate community building before and after class and will be available to activate local emergency medical services in the unlikely event that the need arises. Classes are 75 minutes in duration and meet two times per week.
  Arms: Waitlisted for 8-Week Yoga Class

SUMMARY:
The overall purpose of this study is to adapt a 12-week, standardized in-home yoga program into an 8-week in-home program with a high degree of fidelity, participant adherence, and safety. The Yoga for Seniors program was previously implemented in five rural WI communities with five yoga teachers providing the in-class guidance and support for the standardized program. The investigators seek to convert the program to a telehealth-based approach and deliver the intervention with fidelity to the program, in a safe and effective manner to 120 participants.

DETAILED DESCRIPTION:
Participants will be randomly assigned to immediately begin an 8-week yoga class or complete an 8-week wait (wait-list control). Investigators will examine the measures of interest at pretest (wait-list only), baseline, and posttest to see what, if any, changes are observed after completion of the program. All assessment data collections sessions will be conducted on-line.

Phone screen: All interested participants will complete a phone screen to assess inclusion and exclusion factor for the study.

Testing Procedures: All participants who meet study requirements will complete approximately 60 to 90 minutes of on-line assessments and 60-90 minutes of mailed questionnaires at each testing timepoint (pretest, baseline, and posttest). The assessments will consist of demographic information including a health history form, a semi-structured interview, and a series of questionnaires. The following are the specific assessment components for each time point:

A. Intake and review of forms (Initial Visit (Baseline or Pretest ))

1. Consent form
2. Medical history

B. Clinical measures (all visits)

1. Current medication list
2. Falls history and fear of falls questionnaire
3. Canadian Occupational Performance Measure
4. Physical Activity Scale
5. Perceived Stress Scale
6. Loneliness and Social Isolation Scales
7. Social Network Scale

C. Barriers and facilitators assessments (all visits)

1. technology use assessment survey
2. physical activity readiness scale

D. Exit evaluation (posttest only)

All selected assessment tools have been previously investigated and are valid and reliable for their described use.

During the initial visit (pretest or baseline), participants will complete components A-C listed above.

Individuals in the wait-list control group will complete components B and C during their baseline visit (prior to starting yoga, following their 8-week wait)

Posttest assessment Components B-D will be completed at posttest. Posttest data will be collected within 10 days of the participant's last day of the yoga class.

The group that starts immediately will have 2 time-points of data collection (pretest, posttest), the waitlisted group will have 3 time-points of data collection (baseline, pretest, posttest). Individual results will not be shown or discussed with participants.

The yoga program is an in-home, chair-assisted yoga class focused on balance. Each class will be led by a certified yoga teacher who has completed training the the yoga for Seniors Program. Classes will consist of no more than 12 participants. Each class will be attended by a local community member who will facilitate community building before and after class and will be available to activate local emergency medical services in the unlikely event that the need arises. Classes are 75 minutes in duration and meet two times per week.

See also 12-week program called Yoga for Seniors registered to NCT04889131

ELIGIBILITY:
Inclusion Criteria:

* over 60 years of age
* ability to independently ambulate for at least 10 minutes continuously (with or without an assistive device)
* ability to attend the yoga class for all or most of the 8 weeks
* a previous fall, near-fall or identified fear of falling
* internet access
* vision at or corrected to 20/40 or better

Exclusion Criteria:

* known contraindication for exercise (i.e. a medical doctor has told you not to exercise)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Classes Attended (?0 | up to 8 weeks
  Participant adherence will be measured in part by class attendance. They will have twice weekly classes for 8 weeks, or 16 possible classes to attend.
  [from the purpose: The overall purpose of this study is to adapt the 12-week, standardized in-home yoga program into an 8-week in-home program with a high degree of fidelity, participant adherence, and safety. Are fidelity/adherence/safety a primary outcomes?]

SECONDARY OUTCOMES:
Change in Fall Frequency | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  Change in the frequency of falls will be assessed using a forced-choice paradigm: none, once, 2 to 10 times, weekly, or daily over the last 2 weeks, 1 month, and 6 months.
Change in Activities-Specific Balance Confidence Scale (ABC) | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  The ABC Scale measures a fear of falling. It is a 16-item survey where participants rate their level of self-confidence (0-100, where 100 is the highest self-confidence) for each item. The average score is reported.
Change in Mobility Scale Score | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  Participant is asked to rate their level of confidence (1 extreme confidence to - 10 no confidence at all) that they will not fall in each of 10 activities. Mean confidence level is calculated, lower scores indicate increased confidence.
Change in the Canadian Occupational Performance Measures (COPM) | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  The COPM is composed of the following steps: 1) participant identifies occupational performance problems for self-care and productivity, 2) participant rates each issue on a score of 1-10 (higher scores are more important), 3) participant chooses 5 most important problems, 4) participant rates each issue (1-10) for performance and satisfaction, 5) average score for each (performance and satisfaction) are calculated. Final score for each is 1-10 with higher scores better.
Change in Physical Activity Scale Score | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  12 items scored on a 4 point likert scale for a total possible range of scores from 0-36 where higher scores indicate more physical activity.
Change in Perceived Stress Scale Score | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  10 items scored on a 5 point likert scale for a total possible range of scores from 0-40 where higher scores indicate increased perceived stress.
Loneliness and Social Isolation Scale Score | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  26 items scored on a 4 point likert scale for a total possible range of scores from 0-96 where higher scores indicate increased feelings of loneliness and social isolation.
Social Network Scale Score | baseline (or pretest for immediate group), 8 weeks (posttest for immediate group, pretest for waitlist group), 16 weeks (posttest for waitlist group)
  6 items scored on a 6 point likert scale for a total possible range of scores from 0-30 where higher scores indicate larger social network.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Pickett, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Yoga for Seniors - 12 week program — https://clinicaltrials.gov/ct2/show/NCT04889131